CLINICAL TRIAL: NCT02320760
Title: Physical Activity in Prevention and Treatment of Overweight, Central Obesity and the Metabolic Syndrome - a Randomised Controlled Study in Overweight 65 Year Old Women and Men
Brief Title: Physical Activity on Prescription in Overweight Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Mai-Lis Hellénius, Professor, Proffesor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KI65; 04-520/2 (Other: The regional Ethical review board in Stockholm)
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Low Physical Activity Level; Central Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity, Abdominal; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Physical activity on prescription (Experimental)
  Interventions: Behavioral: Physical activity on prescription
- Ordinary care (No Intervention)

INTERVENTIONS:
Behavioral: Physical activity on prescription
  Arms: Physical activity on prescription

SUMMARY:
This randomized controlled study evaluates the effect of individualized physical activity on prescription (PAP) in older overweight adults. The primary hypothesis is that an individualized prescription of physical activity increases physical activity level in overweight older adults after 6 months. Secondary hypothesis are that the increased physical activity level will improve cardio metabolic risk factors and quality of life.

200 women and men, aged 65 with low physical activity level, overweight, and abdominal obesity, will be randomized to an intervention group or a control group. The control group receives general information about physical activity and registration of physical activity level for one week. The intervention group receives in addition an individualized physical activity on prescription with patient-centered counseling.

After six months both groups go through the same health check-up as at baseline and follow-ups take place after 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 40
* waist circumference over 88 cm for women and 102 cm for men
* basically healthy
* mostly sedentary in their leisure time

Exclusion Criteria:

* current heart disease
* tablet or insulin treated diabetes type 2
* cancer
* other chronic serious illness

Ages: 65 Years to 69 Years | Sex: All
Age Groups: Older Adult
Enrollment: 102 (Actual)
Dates: Start 2005-01; Primary Completion 2007-01 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
physical activity level | 6 months

SECONDARY OUTCOMES:
cardiometabolic risk factors | 6 months

OTHER OUTCOMES:
Quality of life | 6 months

REFERENCES:
- [Derived] Olsson SJ, Borjesson M, Ekblom-Bak E, Hemmingsson E, Hellenius ML, Kallings LV. Effects of the Swedish physical activity on prescription model on health-related quality of life in overweight older adults: a randomised controlled trial. BMC Public Health. 2015 Jul 21;15:687. doi: 10.1186/s12889-015-2036-3. PMID 26193882